CLINICAL TRIAL: NCT04069611
Title: Non Surgical Therapy of Periodontitis in Diabetes Patients: the Adjunctive Use of Probiotics
Acronym: ProDiabet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Sunstar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19/101-R_X
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Diabetes; Periodontitis
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis | interventions — Probiotics; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): Subjects in the test group will receive scaling and root planing, plus the take two probiotic lozenges per day for 3 months (one in the morning and one in the afternoon after brushing their teeth), starting after the last session of SRP. Lozenges will contain L. reuteri (2 x 108 colony forming units/tablet of strains ATCC 55730 and ATCC PTA 5289; Sunstar GUM Periobalance).
  Interventions: Other: Probiotic; Procedure: Scaling and root planing
- Control Group (Placebo Comparator): Subjects assigned to the placebo group will receive scaling and root planing, and will take lozenges exactly like the test ones but without bacteria.
  Interventions: Other: Placebo; Procedure: Scaling and root planing

INTERVENTIONS:
Other: Probiotic — Subjects in the test group will take two probiotic lozenges per day for 3 months (one in the morning and one in the afternoon after brushing their teeth), starting after the last session of SRP. Lozenges will contain L. reuteri (2 x 108 colony forming units/tablet of strains ATCC 55730 and ATCC PTA 5289; Sunstar GUM Periobalance).
  Arms: Test Group
Other: Placebo — Subjects assigned to the placebo group will take lozenges exactly like the test ones but without bacteria.
  Arms: Control Group
Procedure: Scaling and root planing — Mechanical debridement with US and curettes of hard and soft plaque deposits
  Other Names: SRP

SUMMARY:
The aim of this study is to evaluate the clinical and microbiological performance of a probiotic formulation (Sunstar GUM Periobalance) as adjunctive to non-surgical periodontal therapy in patients with diabetes. The null hypothesis is that the adjunctive use of this probiotic formulation would not have any additional benefit over scaling and root planning in the number of residual pockets or in the microbiological impact of the treatment. Conversely, the alternative hypothesis is that the adjunctive use of this formulation would improve the clinical results of non-surgical periodontal therapy when compared to scaling and root planing alone, through a modification of the subgingival biofilm composition.

DETAILED DESCRIPTION:
Diabetes patients will be consecutively selected among those attending the Faculty of Odontology, University Complutense (Madrid, Spain). Patients fulfilling the required criteria will be invited to participate in the study, will be informed on the study purposes, and will be invited to sign and IRB approved informed consent.The study will be designed as a doubled-blind, placebo controlled, parallel, randomized clinical trial with a 6-month follow-up. The patients will be examined for clinical parameters and microbiological sampling, and randomised into two different groups.The following study visits will be scheduled:

Screening visit Potential patient eligibility will be based on the inclusion/exclusion criteria already presented. Patients will be informed about their periodontal condition and treatment needs. Patients willing to participate in the study will be given additional information about the study and upon signing a consent form, they will be appointed for the graduate clinic of Periodontology.

Baseline visit Patients will undergo a comprehensive oral and periodontal examination. Full-mouth clinical measurements of PPD and clinical attachment level (CAL) will be taken at 6 sites per tooth, excluding third molars, and will be rounded to the nearest millimetre using a UNC-15 probe (Hu-Friedy, Chicago, IL, USA). Panoramic radiographs and/or full-mouth periapical radiographs will also be taken, as standard procedures of the postgraduate clinic. Microbiological samples will be taken. The patient smoking history will be recorded and participants will be categorized as: current smokers (those who smoked at least one cigarette per day); never smokers (those who had never smoked in their life); and former smokers (those who had stopped smoking at least 1 year previously). Other relevant aspects of the medical history will be also collected, including the evaluation of the glycated haemoglobin (HbA1c) levels by means of standard laboratory procedures.

Treatment visits Subjects will receive non-surgical periodontal therapy in the form of full-mouth SRP, in two consecutive days, in combination with 0.12% chlorhexidine (Gum Chlorhexidine Oral Rinse, Etoy, Switzerland) application by means of rinsing prior to and at the end of each SRP session. All patients will receive standardized oral hygiene instructions, including the use of a manual toothbrush (GUM® Activital Toothbrush), and interdental brushers (GUM® Trav-ler and GUM® Soft Picks). Instructions will be periodically reinforced.

Immediately after oral hygiene instructions, patients will be randomly allocated to the test or control groups. One investigator before patient recruitment will generate the randomization sequence by blocks. Random assignment into two groups will be carried out with the use of a computer program. Containers will be designed to maintain examiner blinding. The patients will be randomly allocated, with the help of a computer, in two groups:

* Test group: Subjects in the test group will take two probiotic lozenges per day for 3 months (one in the morning and one in the afternoon after brushing their teeth), starting after the last session of SRP. Lozenges will contain L. reuteri (2 x 108 colony forming units/tablet of strains ATCC 55730 and ATCC PTA 5289; Sunstar GUM Periobalance).
* Placebo group: Subjects assigned to the placebo group will take lozenges exactly like the test ones but without bacteria.

Follow up visits after 3 and 6 months Follow up visits will have the objective to monitor the clinical and microbiological changes in the periodontal condition and to evaluate the bacterial re-colonization pattern in the subgingival niche. This phase will include two recall visits, at which clinical measurements will be repeated and microbiological samples will be collected. Oral hygiene will be reinforced. Glycated haemoglobin levels will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed diabetes, for at least 1 year.
* Presence of a minimum of 18 teeth.
* Untreated stages II and III periodontitis with radiographic evidence of generalized alveolar bone loss higher than 30%, and presence of at least one pocket with probing pocket depth (PPD) higher than 5 mm per quadrant with bleeding on probing (BOP).

Exclusion Criteria:

* Subgingival instrumentation within 12 months before baseline examination.
* Use of antibiotics in the three months prior to the study.
* Use of other probiotic products in the month prior the study.
* Systemic diseases that could affect the course of periodontitis or its treatment such as immunological disorders, excluding diabetes.
* Ongoing drug therapy influencing the evaluated clinical parameters (non-steroid inflammatory drugs, etc.).
* Compromised medical conditions requiring prophylactic antibiotic therapy (e.g. patients with valvular prostheses, patients with previous history of bacterial endocarditis, congenital heart diseases like shunts or heart transplant recipients who developed valvular heart disease)
* Pregnancy.
* Stage IV periodontitis, or acute periodontal conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Probing Pocket Depth (PPD) | Baseline, 3 and 6 months
  Change in Probing Pocket Depth (PPD)

SECONDARY OUTCOMES:
Residual Pockets (PPD>4m ) | Baseline, 3 and 6 months
  Percentage of residual pockets
Bleeding on Probing (BOP) | Baseline, 3 and 6 months
  Changes in bleeding on probing
Patient Satisfaction | Baseline, 3 and 6 months
  Patient satisfaction as determined by visual analogue scales (min:0; max:10; 0 indicates worst patient satisfaction, while 10 indicates maximum satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Odontology, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bujaldon R, Montero E, Gamonal JD, Abuelo A, Marin MJ, Iniesta M, Sanz M, Herrera D. Use of the Probiotic Limosilactobacillus reuteri as an Adjunct to Subgingival Instrumentation in the Treatment of Periodontitis Patients With Diabetes: A Randomised Clinical Trial. J Clin Periodontol. 2026 Jan;53(1):26-36. doi: 10.1111/jcpe.70035. Epub 2025 Sep 17. PMID 40958659